CLINICAL TRIAL: NCT07221877
Title: A 12-month Open-label, Phase 4 Multicenter Safety Study to Evaluate the Effect of KarXT on Voiding Dynamics and Urological Safety
Brief Title: A Study to Evaluate the Effect of KarXT on Urological Safety
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN012-0068
Record Dates: First submitted 2025-10-13; First posted 2025-10-28 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KarXT (Experimental)
  Interventions: Drug: Xanomeline/trospium chloride

INTERVENTIONS:
Drug: Xanomeline/trospium chloride — Specified dose on specified days
  Other Names: KarXT; BMS-986510

SUMMARY:
The purpose of this study is to characterize the effect of KarXT on voiding dynamics and urological safety in participants with DSM-5 schizophrenia.

ELIGIBILITY:
Inclusion Criteria

* Male and Female participants (age 18 to 65 years of age, with a primary diagnosis of schizophrenia based on psychiatric evaluation (DSM-5) and confirmed by MINI (v 7.0.2).
* Participants must have a PANSS total score ≤ 80 and CGI-S score ≤ 4, at screening and baseline, and a BMI ≥18 and ≤ 40 kg/m2.
* Participants must be willing and able to discontinue all antipsychotic medications prior to the baseline visit and be willing and able to comply with protocol requirements.

Exclusion Criteria

* Participants with newly diagnosed schizophrenia, any other DSM-5 disorder diagnosed within the past 12 months, alcohol or drug use disorder within the past 12 months, history/presence of clinically significant disease or disorder that would jeopardize participant safety or validity of study results.
* Participants at risk for suicidal behavior, as well as individuals who are pregnant or breastfeeding, will be excluded from the study.
* Other protocol-defined Inclusion/Exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-21 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in voiding dynamics (Qmax) over time | Up to 12 months
Change from baseline in post-void residual volume (PVR) over time | Up to 12 months

SECONDARY OUTCOMES:
Number of participants with a change from baseline in urinalysis parameters over time | Up to 12 months
Change from baseline in IPSS over time | Up to 12 months
Number of participants with electrocardiogram (ECG) abnormalities | Up to 12 months
Number of participants with vital sign abnormalities | Up to 12 months
Number of participants with Adverse Events (AEs) | Up to 12 months
Number of participants with AEs of Special Interest (AESIs) | Up to 12 months
Number of participants with Serious AEs (SAEs) | Up to 12 months
Number of participants with suicidal ideation or behavior | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (16):
- United States (16):
  - Local Institution - 0017, Little Rock, Arkansas
  - Local Institution - 0007, Bellflower, California
  - Local Institution - 0009, Culver City, California
  - CenExel CNS - Garden Grove, Garden Grove, California
  - Local Institution - 0016, Orange, California
  - Local Institution - 0003, Miami, Florida
  - Local Institution - 0008, Miami, Florida
  - Local Institution - 0004, Stuart, Florida
  - Local Institution - 0005, Chicago, Illinois
  - Local Institution - 0010, Chicago, Illinois
  - Local Institution - 0013, Las Vegas, Nevada
  - Local Institution - 0002, Marlton, New Jersey
  - Local Institution - 0012, New York, New York
  - Local Institution - 0014, Philadelphia, Pennsylvania
  - Local Institution - 0001, Austin, Texas
  - InSite Clinical Research, DeSoto, Texas

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07221877.html